CLINICAL TRIAL: NCT07202845
Title: Early Prediction of Neoadjuvant Chemotherapy Response in Bladder Cancer Using Quantitative Multiparametric MRI
Acronym: mpMRI
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Esam Saad Mohamed Darwish, Lecturer, Assiut University
Other Study IDs: PreIRB-Assiut-URO003
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: MIBC; mpMRI; NAC
Keywords: ultiparametric MRI, mpMRI, Diffusion-Weighted Imaging, DWI
MeSH Terms: conditions — Driving Under the Influence | interventions — Multiparametric Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neoadjuvant Chemotherapy + mpMRI Group: Patients with clinical stage cT2-T4 muscle-invasive bladder cancer receiving standard gemcitabine/cisplatin neoadjuvant chemotherapy. Each patient undergoes three multiparametric MRI scans: at baseline (pre-NAC), 24 hours after the first cisplatin dose, and post-NAC before cystectomy. Imaging biomarkers (K^trans^, Ve, ADC index) are analyzed and correlated with pathological response after radical cystectomy.
  Interventions: Diagnostic Test: Multiparametric Magnetic Resonance Imaging (mpMRI)

INTERVENTIONS:
Diagnostic Test: Multiparametric Magnetic Resonance Imaging (mpMRI) — Multiparametric MRI (mpMRI) performed at three defined timepoints: prior to neoadjuvant chemotherapy (baseline), 24 hours after first cisplatin dose in the first NAC cycle, and after completing NAC but before radical cystectomy. Imaging protocols include T2-weighted imaging, diffusion-weighted imaging (DWI), and dynamic contrast-enhanced imaging (DCE-MRI). Quantitative imaging biomarkers such as K^trans^, Ve, and ADC index are extracted and analyzed to evaluate early treatment response and predict pathological outcomes following chemotherapy.
  Other Names: mpMRI

SUMMARY:
Bladder cancer is a prevalent malignancy globally, with muscle-invasive disease having a five-year survival rate below 50%. Neoadjuvant chemotherapy (NAC) before radical cystectomy has shown efficacy for resectable muscle-invasive bladder cancer (MIBC). However, non-response to NAC can lead to delayed surgery and unnecessary toxicity. Magnetic resonance imaging (MRI), particularly multiparametric MRI (mpMRI) with dynamic contrast-enhanced (DCE) and diffusion-weighted imaging (DWI), offers functional and quantitative biomarkers that may predict NAC response early in treatment.

DETAILED DESCRIPTION:
Bladder cancer is a major global health concern, ranking as the sixth most common malignancy in males and the 17th most common in females, with an estimated annual incidence of approximately 550,000 new cases worldwide. Among these, muscle-invasive bladder cancer (MIBC) accounts for around 20% of diagnoses and is associated with a poor prognosis, with five-year survival rates remaining below 50%.

Muscle invasion is a key negative prognostic factor, likely due to early dissemination of micro-metastatic disease at the time of diagnosis. Despite radical cystectomy (RC) being the standard of care for localized MIBC, nearly 50% of patients with ≥T2 stage disease develop distant metastases within two years following surgery, contributing to high disease-specific mortality.

Multiple randomized Phase III trials have demonstrated a survival benefit for neoadjuvant cisplatin-based combination chemotherapy prior to RC in patients with resectable MIBC (clinical stage cT2-T4aN0M0). However, the benefit is largely restricted to responders, as non-responders may experience delays in definitive surgical management and unnecessary chemotherapy-related toxicity without added survival gain.

Given the variability in treatment response, there is a critical need for early and accurate tools to assess therapeutic efficacy and guide personalized treatment strategies. Early identification of non-responders to neoadjuvant chemotherapy (NAC) could allow for timely modification of the treatment plan, avoiding ineffective therapy and associated morbidity.

Magnetic resonance imaging (MRI), particularly multiparametric MRI (mpMRI), has emerged as a valuable imaging modality for bladder cancer due to its superior soft tissue contrast and ability to characterize tissue microarchitecture. mpMRI protocols that include dynamic contrast-enhanced (DCE) imaging and diffusion-weighted imaging (DWI) have shown promise in assessing tumor vascularity, cellularity, and extracellular space - features that are altered during treatment response.

Recent studies suggest that quantitative mpMRI-derived parameters, including the volume transfer constant (K^trans^), the extracellular extravascular volume fraction (Ve), and the apparent diffusion coefficient (ADC), may serve as early biomarkers for predicting response to NAC. Changes in these parameters after the first chemotherapy cycle could provide early indications of therapeutic efficacy, enabling clinicians to adapt treatment pathways accordingly.

This study aims to prospectively evaluate the predictive value of early mpMRI biomarkers - specifically K^trans^, Ve, and ADC - in assessing treatment response following the first cycle of NAC in patients with muscle-invasive bladder cancer. The overarching goal is to determine whether early changes in these imaging parameters correlate with pathological response at cystectomy. This could lead to a more individualized approach to MIBC management and improve clinical outcomes by minimizing ineffective treatment exposure and optimizing timing of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cT2-T4 urothelial carcinoma of the urinary bladder, according to the TNM classification (8), who give informed, written consent on participation in the study and approve all its requirements.
* Planned to receive cisplatin-based NAC followed by radical cystectomy.
* Willing to undergo three mpMRI scans (baseline, 24h post-initial cisplatin, and post-NAC).

Exclusion Criteria:

* Patients who have received pelvic radiotherapy.
* Severe renal impairment
* Previous open or laparoscopic pelvic surgery.
* Presence of distant metastases at diagnosis.
* Patients with contraindications to MRI.
* Ineligibility to cisplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed, clinically localized muscle-invasive urothelial bladder cancer (cT2-T4aN0M0) who are eligible for neoadjuvant cisplatin-based chemotherapy and radical cystectomy, and can safely undergo multiparametric MRI examinations.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Predictive Value of Early mpMRI Biomarkers for Pathological Response to Neoadjuvant Chemotherapy in MIBC | From baseline to time of radical cystectomy (approximately 8-10 weeks)
  This outcome measures the ability of early changes in quantitative multiparametric MRI (mpMRI) biomarkers-specifically the volume transfer constant (K^trans^), extracellular extravascular volume fraction (Ve), and apparent diffusion coefficient (ADC index)-to predict pathological response (complete or partial) to neoadjuvant cisplatin-based chemotherapy in patients with muscle-invasive bladder cancer (MIBC). Pathological response is assessed at the time of radical cystectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Darwish, Lecturer, Principal Investigator — Urology Department, Faculty of Medicine, Assiut University, Assiut, Egypt
Locations (1):
- Amr E. Darwish, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No